CLINICAL TRIAL: NCT05942599
Title: Phase 1 Study of Base Edited CAR T Cells Against AML: Deep Conditioning Ahead of Allogeneic Stem Cell Transplantation
Brief Title: Base Edited CAR T Cells Against AML: Deep Conditioning Ahead of Allogeneic Stem Cell Transplantation
Acronym: CARAML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18IC13
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Phase 1, open label, non-randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose intravenous infusion of a banded dose of CAR33+ T Cells/Kg BECAR33 (Experimental): Patients will undergo careful screening to confirm that this treatment is appropriate for them. Patients will receive BE CAR-33 before their scheduled bone marrow transplant. Chemotherapy will be given prior to BE CAR-33 infusion to improve the ability of CAR T-cells to establish and grow. Patients will then receive a single infusion of the BE CAR-33 cells and will be closely monitored in hospital for the next 4 weeks. Patient will start chemotherapy for their scheduled bone marrow transplant 28 days after BE-CAR33 infusion unless their disease is progressing. Patients will be monitored on the study for 1 year after transplant and then long term in routine clinics.
  Interventions: Biological: Cryopreserved BE CAR33 T Cells (BE752TBTTBCAR33PBL)

INTERVENTIONS:
Biological: Cryopreserved BE CAR33 T Cells (BE752TBTTBCAR33PBL) — Single-dose intravenous infusion (weight-based dosing) of a banded dose of CAR33+ T cells/kg. BECAR33 Total duration of treatment: 28 days follow up: 12 months
  Other Names: BECAR33

SUMMARY:
In this phase 1 clinical trial, the investigators are testing an experimental medicine in children aged 6 months up to 16 years with acute myeloid leukaemia (AML), which has come back (relapsed). The new product is made from white blood cells (T cells) collected from a healthy donor and changed so they can kill leukaemia cells. These 'ready-made' CAR T cells have been made using a new technique called Base Editing to modify their DNA code and have been given the code name 'BE CAR-33'. This technique allows them to work after chemotherapy and also disarms them to prevent effects against normal cells. The main purpose of this study is to assess the safety of the 'BE CAR-33' therapy and to see if ready-made CAR T cells can get rid of Acute Myeloid Leukaemia ahead of a planned bone marrow transplant that will hopefully prevent the leukaemia from returning.

DETAILED DESCRIPTION:
Who can participate? Patients aged 6 months to 16 years with relapsed acute myeloid leukaemia ahead of a planned bone marrow transplant.

What does the study involve? Patients will undergo careful screening to confirm that this treatment is adequate for them. Chemotherapy will be given prior to BE CAR-33 infusion to improve the ability of T-cells to establish and grow. Patients will then receive a single infusion of the BE CAR-33 cells. They will be closely monitored via blood and bone marrow tests for safety and to check the levels of BE CAR-33 and leukaemia cells. The investigators expect patients to be in hospital for 5 weeks for the BE CAR-33 therapy and the transplant will be scheduled 4 weeks after the end of BE CAR33. Patients will be monitored every month for the first three months and then every 6 months.

What are the possible benefits and risks of participating? Taking part in the study of testing 'ready-made' CAR T cells could help reduce the amount of disease and get the patient into remission before a planned bone marrow transplant. Leukaemia is less likely to come back after a bone marrow transplant if levels in the bone marrow are undetectable. The ready-made CAR T cells are being used to try and improve the chances of successful transplantation. Side effects may include low blood cell counts, infections, cytokine storm (severe immune reaction), graft versus host disease (where the donated cells attack the body) and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age ranging between 6 months and <16 years

Medical and therapeutic criteria

* Relapsed AML ahead of scheduled allogeneic haematopoietic stem cell transplantation (allo-SCT).
* Morphologically confirmed with leukemic blasts in the bone marrow (>5%) or a quantifiable MRD by multiparameter flow cytometry and/or quantitative polymerase chain reaction (>10-4)
* CD33+ leukaemia associated immunophenotype (LAIP) on >95% of blasts
* Eligible and fit for allogeneic hematopoietic stem cells transplantation with suitable donor available
* Estimated life expectancy ≥ 12 weeks
* Lansky (age < 16 years at the time of assent/consent) or performance status ≥ 70;
* Eastern Cooperative Oncology Group ECOG performance status < 2.

Exclusion Criteria:

* Patients/parents unwilling to undergo follow-up for 15 years
* Foreseeable poor compliance to the study procedures
* Evidence of disease progression after cytoreduction
* Uncontrollable CNS leukaemia or neurological symptoms defined as CNS grade 3 (per
* National Comprehensive Cancer Network guidelines)
* Absence of suitable HLA matched or mismatched donor
* Weight < 6kgs
* Presence of donor-specific anti-HLA antibodies directed against BE-CAR33
* GvHD requiring systemic therapy
* Systemic steroid therapy prednisolone >0.5mg/kg/day
* Known hypersensitivity to test materials or related compounds
* Active bacterial, fungal or viral infections not controlled by standard of care anti- microbial or anti-viral treatment. Uncontrolled bacteraemia/ fungaemia is defined as the ongoing detection of bacteria/fungus on blood cultures despite antibiotic or anti-fungal therapy. Uncontrolled viraemia is defined as rising viral loads on two consecutive occasions despite antiviral therapy.
* Risk of pregnancy or non-compliance with contraception (if applicable). Girls of childbearing potential must have been tested negative in a pregnancy test within 14 days prior to inclusion.
* Lactating female participants unwilling to stop breastfeeding
* Prior CAR T cell therapy known to be associated with ≥Grade 3 cytokine release syndrome (CRS) or ≥Grade 3 drug-related CNS toxicity

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and description of adverse events after BE-CAR33 Infusion | 1 Year
  Incidence of grade 3-5 toxicities occurring from infusion up to one year follow-up. Severe Adverse reactions of special interest will be CRS, ICANS, GvHD and VOD. American Society of Bone Marrow transplantation grading scales for CRS/ICANS, National institute of health criteria for GvHD and EBMT criteria for VOD will be applied. Common terminology criteria for adverse event (CTCAE) nomenclature will be used to grade other adverse events.

SECONDARY OUTCOMES:
Number of patients achieving disease remission ahead of allo-SCT | 28 Days
  Remission rate will be assessed by bone marrow and CNS evaluation after 28 days. Disease remission is defined as morphological complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) with MRD by flow and/or PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Qasim, Prof, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No